CLINICAL TRIAL: NCT00668213
Title: Antioxidant Systems and Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Paul Sternberg, Professor & Chairman of Ophthalmology-Associate Dean for Adult Clinical Affairs Chief Medical Officer, Vanderbilt University
Other Study IDs: 060471
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective:

The objective of this study was to determine whether the antioxidant supplements used in AREDS shifted the plasma pool of the AREDS subjects to a more reduced state. The AREDS subjects were randomly assigned to one of four treatment groups:

1. antioxidants (500mg Vitamin C, 4000IU Vitamin E, 15mg beta carotene)
2. zinc (80mg zinc oxide, 2mg cupric oxide)
3. antioxidants plus zinc;
4. placebo.

None of the subjects received supplemental GSH or cyst (e) ine.

Age-related macular degeneration (AMD) is the leading cause of severe visual impairment in elderly Americans, with an estimated 15 million people having some form of this disease. AMD primarily affects the central vision and many patients develop severe visual handicaps.

Currently there are no clear established understandings of the etiology or pathogenesis of this disease.

DETAILED DESCRIPTION:
Inclusion Criteria

* Age 55-80
* 70 Participants with Intermediate or Advanced AMD
* 70 participants with no ocular signs of AMD
* Willing to give written informed consent, make the required study visits, and follow instructions
* Any race and either sex

Exclusion Criteria

* Current history of a medical condition that would preclude scheduled study visits or completion of the study (e.g., unstable cardiovascular disease, unstable pulmonary disease, chronic hepatitis, or AIDS).
* Current or history of an ophthalmic disease in the study eye (other than AMD) that would likely compromise or during follow-up could likely compromise the visual acuity of the study eye (e.g., amblyopia, uncontrolled glaucoma with an IOP > 30mmHg, ischemic optic neuropathy, proliferative diabetic retinopathy, clinically relevant nonproliferative diabetic retinopathy, clinically relevant diabetic macular edema, significant active uveitis).
* Clinical signs of myopic retinopathy, or a refraction of > -8 diopter power in current prescription
* Aphakic or psuedophakic patients may be enrolled if there is no funduscopic evidence of degenerative myopia present and if there is no medical history prior to the patient's cataract surgery of either myopic retinopathy or a refraction of > -8 diopters.
* Intraocular surgery in study eye (eye to be treated) within 60 days prior to enrollment
* Presence of a scleral buckle in the study eye
* Currently participating or has participated in a clinical trial that utilized an investigational drug or treatment within 30 days prior to administration of study medication. Daily vitamins and/or mineral therapy are allowed.
* Known medical history of allergy or sensitivity to any component of the drug formulation and/or fluorescein dye that is clinically significant in the investigator's opinion.
* Patient is on oral anticoagulant therapy of Coumadin

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80
* 70 Participants with Intermediate or Advanced AMD
* 70 participants with no ocular signs of AMD
* Willing to give written informed consent, make the required study visits, and follow instructions
* Any race and either sex

Exclusion Criteria:

* Current history of a medical condition that would preclude scheduled study visits or completion of the study (e.g., unstable cardiovascular disease, unstable pulmonary disease, chronic hepatitis, or AIDS).
* Current or history of an ophthalmic disease in the study eye (other than AMD) that would likely compromise or during follow-up could likely compromise the visual acuity of the study eye (e.g., amblyopia, uncontrolled glaucoma with an IOP > 30mmHg, ischemic optic neuropathy, proliferative diabetic retinopathy, clinically relevant nonproliferative diabetic retinopathy, clinically relevant diabetic macular edema, significant active uveitis).
* Clinical signs of myopic retinopathy, or a refraction of > -8 diopter power in current prescription
* Aphakic or psuedophakic patients may be enrolled if there is no funduscopic evidence of degenerative myopia present and if there is no medical history prior to the patient's cataract surgery of either myopic retinopathy or a refraction of > -8 diopters.
* Intraocular surgery in study eye (eye to be treated) within 60 days prior to enrollment
* Presence of a scleral buckle in the study eye
* Currently participating or has participated in a clinical trial that utilized an investigational drug or treatment within 30 days prior to administration of study medication. Daily vitamins and/or mineral therapy are allowed.
* Known medical history of allergy or sensitivity to any component of the drug formulation and/or fluorescein dye that is clinically significant in the investigator's opinion.
* Patient is on oral anticoagulant therapy of Coumadin

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects at risk of macular degeneration
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2006-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to find out if there are changes in the blood that would make you at risk for having age related macular degeneration. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sternberg, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Brantley MA Jr, Osborn MP, Sanders BJ, Rezaei KA, Lu P, Li C, Milne GL, Cai J, Sternberg P Jr. The short-term effects of antioxidant and zinc supplements on oxidative stress biomarker levels in plasma: a pilot investigation. Am J Ophthalmol. 2012 Jun;153(6):1104-9.e2. doi: 10.1016/j.ajo.2011.12.010. Epub 2012 Mar 3. PMID 22381365